CLINICAL TRIAL: NCT07210697
Title: Orthodontic Pain Alleviation With Chewing Gum
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Peter Ngan, Department Chair, Orthodontics, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2506181765
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Orthodontic Appliances
Keywords: Orthodontic Pain; xylitol gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xylitol Gum (Active Comparator): Chew one serving or two pieces of xylitol gum three times per day for a total of six grams of xylitol per day.
  Interventions: Drug: Xylitol Gum
- No Gum (No Intervention): Control group that will refrain from chewing gum.

INTERVENTIONS:
Drug: Xylitol Gum — 1 gram of xylitol per piece of gum with one serving being 2 pieces of gum
  Arms: Xylitol Gum

SUMMARY:
The aim of this study is to determine whether chewing gum can alleviate orthodontic treatment discomfort and improve orthodontic treatment experience. The long-term goal is to enable clinicians to decide whether prescription of chewing gum at the placement of orthodontic appliances can improve patient experience with orthodontic treatment. In specific, a total of 60 patients under the age of 18 will be recruited for the study. Consent will be signed by both the child patient and the parents. 30 patients will be asked to chew xylitol gum and the other 30 patients will refrain from chewing gum and serve as the control group. At the appointment for insertion of orthodontic appliances, patients will be instructed to chew one serving or two pieces of xylitol gum three times per day for a total of six grams of xylitol per day. Patients will participate in a survey at the following timepoints- 4 hours, 24 hours, 48 hours and 7 days. The expectation is that this study will determine the effectiveness of using xylitol to decrease pain in orthodontic patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant and Parents able to sign and understand consent
* Ability to chew gum

Exclusion Criteria:

* Pregnant or Breastfeeding women

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale Baseline | Baseline
  Assessment of pain on a visual analogue scale with the scale being 0= very comfortable and 10= severe discomfort with 10 being the worst outcome.
Visual analogue scale 4 hours post treatment | 4 hours post treatment
  Assessment of pain on a visual analogue scale with the scale being 0= very comfortable and 10= severe discomfort with 10 being the worst outcome.
Visual analogue scale 24 hours post treatment | 24 hours post treatment
  Assessment of pain on a visual analogue scale with the scale being 0= very comfortable and 10= severe discomfort with 10 being the worst outcome.
Visual analogue scale 48 hours post treatment | 48 hours post treatment
  Assessment of pain on a visual analogue scale with the scale being 0= very comfortable and 10= severe discomfort with 10 being the worst outcome.
Visual analogue scale 1 week post treatment | 1 week post treatment
  Assessment of pain on a visual analogue scale with the scale being 0= very comfortable and 10= severe discomfort with 10 being the worst outcome.
Comfort Level for Biting Baseline | Baseline
  Measured using the question "Select the level of comfort you have concerning biting." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Biting 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select the level of comfort you have concerning biting." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Biting 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select the level of comfort you have concerning biting." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Biting 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select the level of comfort you have concerning biting." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Biting 1 week post treatment | 1 week post treatment
  Measured using the question "Select the level of comfort you have concerning biting." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Chewing Baseline | Baseline
  Measured using the question "Select the level of comfort you have concerning chewing." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Chewing 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select the level of comfort you have concerning chewing." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Chewing 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select the level of comfort you have concerning chewing." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Chewing 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select the level of comfort you have concerning chewing." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Chewing 1 week post treatment | 1 week post treatment
  Measured using the question "Select the level of comfort you have concerning chewing." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Fitting Back Teeth Baseline | Baseline
  Measured using the question "Select the level of comfort you have concerning fitting your back teeth together." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Fitting Back Teeth 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select the level of comfort you have concerning fitting your back teeth together." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Fitting Back Teeth 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select the level of comfort you have concerning fitting your back teeth together." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Fitting Back Teeth 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select the level of comfort you have concerning fitting your back teeth together." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Fitting Back Teeth 1 week post treatment | 1 week post treatment
  Measured using the question "Select the level of comfort you have concerning fitting your back teeth together." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Fitting Front Teeth Baseline | Baseline
  Measured using the question "Select the level of comfort you have concerning fitting your front teeth together." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Fitting Front Teeth 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select the level of comfort you have concerning fitting your front teeth together." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Fitting Front Teeth 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select the level of comfort you have concerning fitting your front teeth together." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Fitting Front Teeth 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select the level of comfort you have concerning fitting your front teeth together." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Fitting Front Teeth 1 week post treatment | 1 week post treatment
  Measured using the question "Select the level of comfort you have concerning fitting your front teeth together." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Speech Baseline | Baseline
  Measured using the question "Select the level of comfort you have concerning speech." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Speech 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select the level of comfort you have concerning speech." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Speech 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select the level of comfort you have concerning speech." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Speech 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select the level of comfort you have concerning speech." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for Speech 1 week post treatment | 1 week post treatment
  Measured using the question "Select the level of comfort you have concerning speech." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for popping and clicking of the jaw joint Baseline | Baseline
  Measured using the question "Select the level of comfort you have concerning popping and clicking of the jaw joint." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for popping and clicking of the jaw joint 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select the level of comfort you have concerning popping and clicking of the jaw joint." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for popping and clicking of the jaw joint 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select the level of comfort you have concerning popping and clicking of the jaw joint." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for popping and clicking of the jaw joint 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select the level of comfort you have concerning popping and clicking of the jaw joint." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Comfort Level for popping and clicking of the jaw joint 1 week post treatment | 1 week post treatment
  Measured using the question "Select the level of comfort you have concerning popping and clicking of the jaw joint." using a Likert type scale of 0-10 [very comfortable (0) to mild discomfort (5) to severely uncomfortable (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with appearance of teeth Baseline | Baseline
  Measured using the question "Select how you feel about the appearance of your teeth" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with appearance of teeth 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select how you feel about the appearance of your teeth" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with appearance of teeth 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select how you feel about the appearance of your teeth" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with appearance of teeth 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select how you feel about the appearance of your teeth" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with appearance of teeth 1 week post treatment | 1 week post treatment
  Measured using the question "Select how you feel about the appearance of your teeth" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with appearance of facial profile Baseline | Baseline
  Measured using the question "Select how you feel about your facial profile" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with appearance of facial profile 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select how you feel about your facial profile" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with appearance of facial profile 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select how you feel about your facial profile" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with appearance of facial profile 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select how you feel about your facial profile" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with appearance of facial profile 1 week post treatment | 1 week post treatment
  Measured using the question "Select how you feel about your facial profile" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with general appearance of face Baseline | Baseline
  Measured using the question "Select how you feel about the general appearance of your face" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with general appearance of face 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select how you feel about the general appearance of your face" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with general appearance of face 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select how you feel about the general appearance of your face" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with general appearance of face 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select how you feel about the general appearance of your face" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with general appearance of face 1 week post treatment | 1 week post treatment
  Measured using the question "Select how you feel about the general appearance of your face" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with overall appearance Baseline | Baseline
  Measured using the question "Select how you feel about your overall appearance" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with overall appearance 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select how you feel about your overall appearance" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with overall appearance 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select how you feel about your overall appearance" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with overall appearance 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select how you feel about your overall appearance" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with overall appearance 1 week post treatment | 1 week post treatment
  Measured using the question "Select how you feel about your overall appearance" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with general health Baseline | Baseline
  Measured using the question "Select how you feel about your general health" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with general health 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select how you feel about your general health" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with general health 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select how you feel about your general health" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with general health 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select how you feel about your general health" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with general health 1 week post treatment | 1 week post treatment
  Measured using the question "Select how you feel about your general health" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with self-esteem Baseline | Baseline
  Measured using the question "Select how you feel about your self-esteem" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with self-esteem 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select how you feel about your self-esteem" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with self-esteem 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select how you feel about your self-esteem" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with self-esteem 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select how you feel about your self-esteem" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with self-esteem 1 week post treatment | 1 week post treatment
  Measured using the question "Select how you feel about your self-esteem" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with socializing Baseline | Baseline
  Measured using the question "Select how comfortable you feel about socializing with peers" using a Likert type scale of 0-10 [confident in socializing (0) to neutral (5) to avoid socializing (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with socializing 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select how comfortable you feel about socializing with peers" using a Likert type scale of 0-10 [confident in socializing (0) to neutral (5) to avoid socializing (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with socializing 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select how comfortable you feel about socializing with peers" using a Likert type scale of 0-10 [confident in socializing (0) to neutral (5) to avoid socializing (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with socializing 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select how comfortable you feel about socializing with peers" using a Likert type scale of 0-10 [confident in socializing (0) to neutral (5) to avoid socializing (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with socializing 1 week post treatment | 1 week post treatment
  Measured using the question "Select how comfortable you feel about socializing with peers" using a Likert type scale of 0-10 [confident in socializing (0) to neutral (5) to avoid socializing (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with school performance Baseline | Baseline
  Measured using the question "Select how you feel about your performance in school" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with school performance 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select how you feel about your performance in school" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with school performance 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select how you feel about your performance in school" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with school performance 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select how you feel about your performance in school" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with school performance 1 week post treatment | 1 week post treatment
  Measured using the question "Select how you feel about your performance in school" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with being out in public Baseline | Baseline
  Measured using the question "Select how you feel about being out in public" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with being out in public 4 hours post treatment | 4 hours post treatment
  Measured using the question "Select how you feel about being out in public" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with being out in public 24 hours post treatment | 24 hours post treatment
  Measured using the question "Select how you feel about being out in public" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with being out in public 48 hours post treatment | 48 hours post treatment
  Measured using the question "Select how you feel about being out in public" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Satisfaction with being out in public 1 week post treatment | 1 week post treatment
  Measured using the question "Select how you feel about being out in public" using a Likert type scale of 0-10 [very good (0) to neutral (5) to very bad (10)] with 0 being the best outcome and 10 being the worst.
Self-Reported Level of Neuroticism Baseline | Baseline
  Measured using the question "How do you fall on a scale of neuroticism?" Investigators provide the definition of neuroticism as the following: Neuroticism is a tendency to experience emotions such as anxiety, depression, and anger. The scale used is a Likert type scale with 0= Very Neurotic, 5= Somewhat Neurotic, and 10= Not Neurotic. Higher scores indicate lower levels of neuroticism.
Self-Reported Introversion/extroversion Baseline | Baseline
  Measured using the question "How do you fall on a scale of introversion/extroversion?" Investigators provide the definition of neuroticism as the following: Introvert is someone who is socially reserved; Ambivert falls in the middle; Extrovert is someone who is very socially outgoing. The scale used is a Likert type scale with 0= Introvert, 5= Ambivert, and 10= Extrovert. Higher scores indicate higher levels of being socially outgoing.
Adherence to chewing gum instructions 4 hours post treatment | 4 hours post treatment
  Percentage of participants that adhered to the instructions of not chewing gum. Measured using the yes/no question "Did you follow the instructions about chewing gum?" Responses are binary: Yes or No. A response of "Yes" indicates adherence to the chewing gum instructions.
Adherence to chewing gum instructions 24 hours post treatment | 24 hours post treatment
  Percentage of participants that adhered to the instructions of not chewing gum. Measured using the yes/no question "Did you follow the instructions about chewing gum?" Responses are binary: Yes or No. A response of "Yes" indicates adherence to the chewing gum instructions.
Adherence to chewing gum instructions 48 hours post treatment | 48 hours post treatment
  Percentage of participants that adhered to the instructions of not chewing gum. Measured using the yes/no question "Did you follow the instructions about chewing gum?" Responses are binary: Yes or No. A response of "Yes" indicates adherence to the chewing gum instructions.
Adherence to chewing gum instructions 1 week post treatment | 1 week post treatment
  Percentage of participants that adhered to the instructions of not chewing gum. Measured using the yes/no question "Did you follow the instructions about chewing gum?" Responses are binary: Yes or No. A response of "Yes" indicates adherence to the chewing gum instructions.
Adherence to avoiding pain medications instructions 4 hours post treatment | 4 hours post treatment
  Percentage of participants that adhered to the instructions of avoiding pain medication. Measured using the yes/no question "Did you follow the instructions about avoiding pain medications such as Tylenol or Advil?" Responses are binary: Yes or No. A response of "Yes" indicates adherence to the avoiding pain medications instructions.
Adherence to avoiding pain medications instructions 24 hours post treatment | 24 hours post treatment
  Percentage of participants that adhered to the instructions of avoiding pain medication. Measured using the yes/no question "Did you follow the instructions about avoiding pain medications such as Tylenol or Advil?" Responses are binary: Yes or No. A response of "Yes" indicates adherence to the avoiding pain medications instructions.
Adherence to avoiding pain medications instructions 48 hours post treatment | 48 hours post treatment
  Percentage of participants that adhered to the instructions of avoiding pain medication. Measured using the yes/no question "Did you follow the instructions about avoiding pain medications such as Tylenol or Advil?" Responses are binary: Yes or No. A response of "Yes" indicates adherence to the avoiding pain medications instructions.
Adherence to avoiding pain medications instructions 1 week post treatment | 1 week post treatment
  Percentage of participants that adhered to the instructions of avoiding pain medication. Measured using the yes/no question "Did you follow the instructions about avoiding pain medications such as Tylenol or Advil?" Responses are binary: Yes or No. A response of "Yes" indicates adherence to the avoiding pain medications instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ngan, DMD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No